CLINICAL TRIAL: NCT07168291
Title: The Safety and Efficacy of Novel Bispecific AbTCR (Anti-CD19/CD22)-T Cells in Patients With Relapsed or Refractory B-cell Lymphoma: An Open-label, Single-arm Clinical Study
Brief Title: Novel Bispecific AbTCR (Anti-CD19/CD22)-T Cells in Relapsed or Refractory B-cell Lymphoma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Eureka Therapeutics Inc. (Industry)
Responsible Party: Principal Investigator, He Pengcheng, Professor, First Affiliated Hospital Xi'an Jiaotong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2025LSYY-461
Record Dates: First submitted 2025-09-05; First posted 2025-09-11 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL); Follicular Lymphoma ( FL); Burkitt Lymphoma
Keywords: AbTCR-T; CD19/CD22; B-cell lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Burkitt Lymphoma; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conditioning chemotherapy plus AbTCR (anti-CD19/CD22)-T cells (Experimental): The trial will enroll 3 patients with relapsed or refractory B-cell lymphoma.
  Interventions: Drug: Conditioning chemotherapy followed by AbTCR (anti-CD19/CD22)-T cell infusion

INTERVENTIONS:
Drug: Conditioning chemotherapy followed by AbTCR (anti-CD19/CD22)-T cell infusion — Cyclophosphamide 250 mg/m2 and fludarabine 30 mg/m2 IV infusion on day -5, -4, and -3. AbTCR (anti-CD19/CD22)-T cell IV infusion on day 0.

SUMMARY:
This is an open-lable, single arm, non-randomized study to evaluate the primary safety and efficacy of the novel bispecific AbTCR (anti-CD19/CD22)-T cells in patients with relapsed or refractory B-cell lymphoma

DETAILED DESCRIPTION:
The investigators previously developed CD19-targeted ET019003 T cells by fusing the Fab fragment with γ/δ TCR constant chain plus adding a co-stimulatory molecule. Among 12 treated patients enrolled in the phase I clinical trial (NCT03642496), 6 achieved complete remission and no serious adverse events were observed, demonstrating that ET019003 T cells are both safe and effective. However, its efficacy is limited in patients with loss of CD19 expression. To overcome tumor immune escape driven by antigen loss, investigators designed the novel AbTCR-T cells simultaneously targeting CD19 and CD22. This trial is conducted to explore the safety and efficacy of AbTCR (anti-CD19/CD22)-T cells in treating patients with refractory/relapsed aggressive lymphomas.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 18 years;
2. Pathologically diagnosed CD19+/CD22+ B-cell lymphoma;
3. Relapsed or refractory after at least two prior lines of therapy;
4. Patient's main organs functioning well:

   1. Cardiac function: Left ventricular ejection fraction ≥50%;
   2. Liver function: ALT and AST ≤2.5 × upper limit of normal (ULN), total bilirubin ≤2 × ULN;
   3. Renal function: Serum creatinine ≤3.0 mg/dL (≤260 μmol/L);
   4. Pulmonary function: ≤CTCAE grade 1 dyspnea and Indoor oxygen saturation ≥92%;
   5. Adequate bone marrow function as assessed by the investigator to receive lymphodepleting chemotherapy;
5. Adequate vascular access for leukapheresis;
6. Women of childbearing potential (all women physiologically capable of becoming pregnant) must agree to use highly effective contraception for 1 year after AbTCR (anti-CD19/CD22)-T cell infusion, such as copper-containing intrauterine device, hormonal implants, or tubal ligation; male subjects with partners of childbearing potential must agree to use effective barrier contraception for 1 year after AbTCR (anti-CD19/CD22)-T cell infusion;
7. Patient or his or her legal guardian voluntarily participates in and signs an informed consent form.

Exclusion Criteria:

1. Lymphoma involving only the central nervous system (CNS), or secondary CNS lymphoma patients judged by the investigator to be at high risk for AbTCR (anti-CD19/CD22)-T cell therapy;
2. History of other malignancies not in complete remission for at least 2 years (the following conditions are exempt from the 2-year restriction: non-melanoma skin cancer, completely resected stage I tumors with low risk of recurrence, treated localized prostate cancer, biopsy-confirmed cervical carcinoma in situ, or PAP smear showing squamous intraepithelial lesion);
3. Any of the following at screening:

   1. Positive hepatitis B surface antigen (HBsAg) (regardless of hepatitis B virus DNA copy number);
   2. Positive hepatitis B core antibody (HBcAb) with increased hepatitis B virus DNA copy number;
   3. Hepatitis C, human immunodeficiency virus (HIV), or syphilis infection;
4. Deep vein thrombosis (DVT) or pulmonary embolism (PE) within 3 months prior to signing informed consent;
5. Ongoing anticoagulant therapy for deep vein thrombosis (DVT) or pulmonary embolism (PE) within 3 months prior to signing informed consent;
6. Uncontrolled systemic fungal, bacterial, viral, or other infection;
7. Acute or chronic graft-versus-host disease (GvHD);
8. History of any of the following cardiovascular diseases within the past 6 months: Class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant heart disease;
9. History of or current clinically significant CNS disease at screening, such as epilepsy, seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychiatric illness;
10. Pregnant or breastfeeding women. Women of childbearing potential must have a negative serum pregnancy test within 48 hours prior to starting lymphodepleting chemotherapy;
11. Use of any of the following drugs or treatments within the specified timeframes prior to leukapheresis:

    1. Alemtuzumab within 6 months prior to leukapheresis;
    2. Cladribine within 3 months prior to leukapheresis;
    3. Fludarabine within 3 months prior to leukapheresis;
    4. Anti-CD20 monoclonal antibody within 7 days prior to leukapheresis;
    5. Venetoclax within 4 days prior to leukapheresis;
    6. Idelalisib within 2 days prior to leukapheresis;
    7. Lenalidomide within 1 day prior to leukapheresis;
    8. Therapeutic doses of corticosteroids (defined as prednisone or equivalent >20 mg/day) within 7 days prior to leukapheresis; physiological replacement, topical, and inhaled steroids are permitted;
    9. Non-lymphocytotoxic chemotherapy within 1 week prior to leukapheresis. Oral chemotherapy drugs are allowed if at least 3 half-lives have passed prior to leukapheresis;
    10. Lymphocytotoxic chemotherapy (e.g., cyclophosphamide, ifosfamide, bendamustine, chlorambucil, or melphalan) within 2 weeks prior to leukapheresis;
    11. Investigational drugs within 4 weeks prior to leukapheresis. However, subjects who had no response or disease progression during experimental treatment and for whom at least 3 half-lives have passed since the last dose prior to leukapheresis are allowed;
    12. GvHD therapy (e.g., calcineurin inhibitors, methotrexate or other chemotherapeutic agents, mycophenolate, rapamycin, thalidomide, immunosuppressive antibodies such as anti-TNF, anti-IL6, or anti-IL6R) within 4 weeks prior to leukapheresis and AbTCR (anti-CD19/CD22)-T cell infusion;
    13. Donor lymphocyte infusion (DLI) within 6 weeks prior to AbTCR (anti-CD19/CD22)-T cell administration;
    14. Radiotherapy within 6 weeks prior to leukapheresis, including large bone marrow areas such as the sternum or pelvis. Patients with progressive disease at irradiated sites or PET-positive lesions at non-irradiated sites are eligible. Radiotherapy to a single site is allowed within 2 weeks prior to leukapheresis if there are PET-positive lesions at other non-irradiated sites;
    15. If prior immunotherapy such as anti-PD1 or anti-PD-L1 was used, at least 5 half-lives must have passed between the last dose and AbTCR (anti-CD19/CD22)-T cell infusion;
12. Prior allogeneic hematopoietic stem cell transplantation;
13. Other conditions considered inappropriate by the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | 3 years
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0) or ASTCT consensus.

SECONDARY OUTCOMES:
Overall response rate (ORR) of administering AbTCR (anti-CD19/CD22)-T cells in relapsed/refractory B cell lymphoma. | 3 years
  ORR will be assessed from AbTCR (anti-CD19/CD22)-T cell infusion to death or last follow-up (censored).
Overall survival (OS) of administering AbTCR (anti-CD19/CD22)-T cells in relapsed/refractory B-cell lymphoma. | 3 years
  OS will be assessed from AbTCR (anti-CD19/CD22)-T cell infusion to death or last follow-up (censored).
Progress-free survival (PFS) of administering AbTCR (anti-CD19/CD22)-T cells in relapsed/refractory B-cell lymphoma. | 3 years
  PFS will be assessed from AbTCR (anti-CD19/CD22)-T cell infusion to death or last follow-up (censored).
Duration of Response (DOR) of administering AbTCR (anti-CD19/CD22)-T cells in relapsed/refractory B-cell lymphoma. | 3 years
  DOR will be assessed from AbTCR (anti-CD19/CD22)-T cell infusion to death or last follow-up (censored).

OTHER OUTCOMES:
Expansion, persistence, and infiltration of AbTCR (anti-CD19/CD22)-T cells in peripheral blood, bone marrow, and tumor tissues. | 3 years
  AbTCR (anti-CD19/CD22)-T cells will be determined by flow cytometry and ddPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Pengcheng He, M.D., Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China